CLINICAL TRIAL: NCT06569784
Title: A Clinical Study on Absorption, Metabolism, and Excretion of [14C]HSK31858 in Healthy Adult Male Chinese Subjects - Mass Balance and Biotransformation of [14C]HSK31858 in Human.
Brief Title: Mass Balance Study of [14C]HSK31858 in Healthy Adult Male Chinese Subjects.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xizang Haisco Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK31858-103
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 40 mg/120 μCi[14C]HSK31858 (Experimental): [14C]HSK31858
  Interventions: Drug: [14C]HSK31858

INTERVENTIONS:
Drug: [14C]HSK31858 — A single oral dose of 40 mg/120 μCi [14C]HSK31858 after fasting for at least 10 hours.

SUMMARY:
This is a single-center, nonrandomized, and open design study to investigate the pharmacokinetics, mass balance, metabolism and excretion of HSK31858 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese male subjects, Age: 18~45 years old (inclusive);
2. Body weight ≥50.0 kg and BMI of 19 to 26 kg/m^2(inclusive);
3. Subjects who voluntarily signed the informed consent form, are able to communicate with the investigator and complete all study procedures as per the protocol.

Exclusion Criteria:

Clinical examination:

1. After physical examination, vital signs, laboratory tests (hematology, blood biochemistry, coagulation, urinalysis, stool analysis + occult blood, thyroid function), ophthalmological examination (slit lamp, intraocular pressure and fundus photography), 12-lead electrocardiogram [Fridericia-corrected QT (QTcF)-interval, which in men should be between 350-450ms (inclusive)], chest X-ray (PA and lateral), and abdominal ultrasound (liver, gallbladder, pancreas, spleen, kidney) are abnormal and clinically significant;
2. Subjects tested positive for hepatitis B surface antigen or E antigen, hepatitis C antibody, combined human immunodeficiency virus antigen/antibody (HIV-Ag/Ab), or Treponema pallidum antibody;

   Medication history:
3. Subjects who have used prescription, over-the-counter, or healthcare drugs, including Western or proprietary Chinese medicines, within 14 days or 5 half-lives of the drug, whichever is longer, prior to screening;
4. Subjects who have articipated in any clinical trial and received test drug or medical device intervention within 3 months prior to screening;
5. Anyone who has used any drug that inhibits or induces CYP3A activity or P-gp inhibitors within 30 days prior to screening;

   Disease history and surgical history:
6. Prior or current history of any clinically serious disease of the cardiovascular, digestive, respiratory, endocrine, neurological, haematological, immunological, dermatological, oncological, psychiatric, and metabolic abnormalities or any other disease or physiological condition capable of interfering with the study results;
7. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsades de pointes, ventricular tachycardia, atrioventricular block, QT prolongation syndrome, or symptoms of QT prolongation syndrome, or a family history of the disease (as evidenced by genetic predisposition or a close relative's sudden death from cardiac causes at a young age);
8. Subjects with a previous diagnosis of periodontitis or/and palmoplantar hyperkeratosis who are screened with the following problems:

   * Subjects with current signs of gingivitis/periodontitis;
   * Subjects with a history of hyperkeratosis of the palms or soles or erythema;
9. Subjects who had major surgery or incompletely healed surgical incisions within 6 months prior to the screening, including, but not limited to, any surgery with significant risk of bleeding, prolonged general anaesthesia or incisional biopsy, or significant traumatic injury (with the exception of healed surgery of appendicitis or prolapse of the anus);
10. Subjects with hyperactive immune response, including: clear sensitive to DPP1 inhibitors or any excipients of the drug in this trial, allergy to two or more other drugs or food ingredients or special dietary requirements and inability to comply with a uniform diet;
11. Comorbidities with haemorrhoids or perianal disease with regular/ongoing blood in stool, irritable bowel syndrome, inflammatory bowel disease;

    Lifestyle habits:
12. Irregular bowel movements or diarrhoea;
13. Alcohol abuse or frequent alcohol drinking within 6 months prior to screening, that is, > 14 units of alcohol consumption per week (1 unit = 360 mL beer or 45 mL of liquor with 40% alcohol or 150 mL wine), or positive result for breath alcohol test at screening;
14. Subjects who smoke more than 5 cigarettes a day or have habitual use of nicotine containing products within 3 months prior to screening and fail to quit smoking during the trial;
15. Subjects with a long history of drug abuse or dependence with a positive urine screen for drug abuse;
16. Subjects with habitual consumption of grapefruit juice or excessive tea (more than 8 cups a day, 1 cup = 250mL), excessive caffeine (more than 3 cups of coffee a day, etc.) that cannot be stopped during the trial;

    Other:
17. Subjects who engage in work requiring long-term exposure to radioactive conditions; or those with significant radioactive exposure within 1 year prior to the trial (≥ 2 chest/abdominal CT, or ≥ 3 other types of X-ray tests); or those who have participated in radiopharmaceutical studies within 1 year;
18. Subjects with a history of fainting during acupuncture or blood phobia, difficulty in collecting blood, or inability to tolerate blood collection by venipuncture;
19. The presence of tattoos or scars on any part of the skin that, in the judgement of the investigator, interfere with the safety assessment;
20. Subjects having a birth plan during the trial and in 1 year after trial completion, or subjects or their spouses who refuse to take rigorous contraceptive measures (including use of condoms, contraceptive sponges, contraceptive gels, contraceptive diaphragms, intrauterine devices, oral or injectable contraceptives, contraceptive implants, etc.) during the trial and in 1 year after trial completion;
21. Subjects who had blood loss or blood donation of up to 400 mL in 3 months prior to screening, or who had received blood transfusion in 1 month prior to screening;
22. Subjects unsuitable for participating in this trial for any other reason as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Total radioactivity ecovery rates in urine | during periods of 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours, 24-48 hours, 48-72 hours, 72-96 hours, 96-120 hours, 120-144 hours, 144-168 hours, 168-192 hours, 192-216 hours, 216-240 hours, 240-264 hours, 264-288 hours, and 288-312 hours post-dose
  Total radioactivity ecovery rates in urine at each time interval.
Total radioactivity ecovery rates in feces | during periods of 0-24 hours, 24-48 hours, 48-72 hours, 72-96 hours, 96-120 hours, 120-144 hours, 144-168 hours, 168-192 hours, 192-216 hours, 216-240 hours, 240-264 hours, 264-288 hours, and 288-312 hours post-dose
  Total radioactivity ecovery rates in feces at each time interval.
Cumulative total radioactivity recovery rates | From the start of administration to 312 hours post-dose
  Cumulative total radioactivity recovery rates of [14C]HSK31858 in excretion (urine and faeces) accounting for total radiation drug dose.
Cmax of total radioactivity | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of total radioactivity in plasma
AUC(0-t) of total radioactivity | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of total radioactivity in plasm
AUC(0-∞) of total radioactivity | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of total radioactivity in plasm
%AUC | From the start of administration to 312 hours post-dose
  Human plasma parent drug and its metabolites as a percentage of total plasma radioactivity exposure
% administered dose | From the start of administration to 312 hours post-dose
  Human urine and feces parent drug and its metabolites as a percentage of administered dose
Identification of the main metabolites | From the start of administration to 312 hours post-dose
  Identification of the main metabolites of HSK31858 in plasma, urine, and feces.

SECONDARY OUTCOMES:
AUC(0-t) | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of the parent drug HSK31858, metabolite M4 and other metabolites (if applicable) in plasma
AUC(0-∞) | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of the parent drug HSK31858, metabolite M4 and other metabolites (if applicable) in plasma
Cmax | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of the parent drug HSK31858, metabolite M4 and other metabolites (if applicable) in plasma
Tmax | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of the parent drug HSK31858, metabolite M4 and other metabolites (if applicable) in plasma
t1/2 | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of the parent drug HSK31858, metabolite M4 and other metabolites (if applicable) in plasma
Mean Residence Time | From the start of administration to 312 hours post-dose
  The pharmacokinetic parameters of the parent drug HSK31858, metabolite M4 and other metabolites (if applicable) in plasma
AEs | From the time of signing ICF to the end of follow-up，up to 14 days.
  The incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China